CLINICAL TRIAL: NCT02361008
Title: TEE-guided Perventricular Device Closure Through Minithoracotomy vs Traditional Surgery Repair Via CBP in Treatment of Infundibular Ventricular Septal Defect：A Two-center Clinical Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial:Treatments on Infundibular Ventricular Septal Defect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bentong Yu (Other)
Collaborators: The Third Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor-Investigator, Bentong Yu, Director of Thoracic and Cardiovascular Surgery Department, The First Affiliated Hospital of Nanchang University
Organization: The First Affiliated Hospital of Nanchang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCQ-2012-80-SXHZJH-1
Record Dates: First submitted 2015-01-29; First posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Heart Septal Defects, Ventricular; Double Outlet Right Ventricle, Noncommitted VSD; Double Outlet Right Ventricle, Subaortic VSD; Double Outlet Right Ventricle, Subpulmonary VSD; Supracristal Ventricular Septal Defect
Keywords: Infundibular Ventricular Septal Defect; occlusion; TEE-guided; asymmetric occluder; surgical repair
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Double Outlet Right Ventricle; Bites and Stings

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- TPDC group (Experimental): Patients who matched inclusion criteria and randomly divided into TPDC group underwent the TEE-guided perventricular device closure without CBP. But of them,who underwent TPDC failure during the procedure would be dropped out of the trial.
  Interventions: Device: TEE-guided perventricular device closure without CBP; Procedure: Surgery repair with CBP
- SR group (Experimental): Patients who matched inclusion criteria and randomly assigned into SR group underwent the surgery repair with CBP.
  Interventions: Procedure: Surgery repair with CBP

INTERVENTIONS:
Device: TEE-guided perventricular device closure without CBP — Perventricular device closure through minithoracotomy under the TEE-guidance without CBP.The device is an eccentric occluder made by Shanghai Shape Memory Alloy Co.,Ltd in Shanghai,China
  Other Names: TPDC
  Arms: TPDC group
Procedure: Surgery repair with CBP — Traditional surgery repair under the CBP.
  Other Names: SR

SUMMARY:
The purpose of this study is to investigate the security and validity of transesophageal echocardiography(TEE)-guided perventricular device closure(TPDC) through minithoracotomy in treatment of infundibular ventricular septal defect(IVSD) with asymmetric occluder.

DETAILED DESCRIPTION:
Ventricular septal defect(VSD) , which accounted for about 20% of all congenital heart defects (CHDs) , is among the most common congenital heart malformations，among which infundibular ventricular septal defects(IVSD) is the least common type(18%）.Multiple names for IVSD are in use. They can also be labeled conal VSD, subpulmonary VSD, subarterial VSD, doubly committed VSD, intracristal VSD，or supracristal VSD. These multiple denominations are not attached to specifically different anatomic subtypes.At present, the main methods to treat the specific anatomic condition contain conventional surgical repair(SR) and transcatheter interventional closure. The former need extracorporeal circulation，thus the side effects of extracorporeal circulation are inevitable，such as on the central nervous system, respiratory system, urinary system, etc. Although the latter has the characteristics of minimally invasive, patients should be exposed in X-ray withstanding potential risk of radiation. On the other hand，there are limits with age for patients who underwent transcatheter closure because of small vessel size. Fully developed blood vessels are to reach a certain diameter, but children need be up to 3 years old or so. In addition,the aortic valve was easily injured by wire and atrioventricular block was reported.Since the surrounding structure is complicated and the defect is too high, device closure of an IVSD is difficult to succeed in transcatheter approach. Traditional repair via cardiopulmonary bypass(CBP) is widely used to treat this kind of diseases. Past decade，with the development of technology and society，TEE-guided surgical occlusion through minithoracotomy was used to treat CHDs in an increasing number of popularity，avoiding the inherent risks of cardiopulmonary bypass and radiation,etc. But it is rarely reported to treat IVSD by minimally invasive perventricular device closure without CBP.

ELIGIBILITY:
Inclusion Criteria:

(1) patients with single IVSD indicated by TTE，without concomitant cardiac malformation, serious arrhythmia or other important non-cardiac diseases；(2) patients whose ventricular septal defects from aortic residual < 3 mm, preoperative without aortic regurgitation or only mild reflux, defect size ≤10 mm;

Exclusion Criteria:

(1) defect size > 10 mm in diameter; （2) Preoperative with above moderate aortic valve prolapse (or) closed incompletely; (3) Eisenmenger syndrome caused by pulmonary hypertension,(4)decide temporarily to change method before surgery;(5) not signed informed consent application

Ages: 7 Days to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20121212 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Surgery success rate | two months
  Surgery success means that patients in both TPDC and SR group don't change their surgery type either undergo a repeat surgery.

SECONDARY OUTCOMES:
Hospitalization costs | 1 months
  The hospitalization costs calculated from hospital admission to hospital discharge

OTHER OUTCOMES:
Length of hospital stay (post-op) | 1 months
  Length of hospital stay refers in particular to the post-op stay in hospital.
Mean bleeding volume | 6 hours
  The mean bleeding volume only referred during the procedure
Volume of drainage | 1 weeks
  The volume of drainage is calculated from being moved off operating table to being pulled out drainage tube.
Procedure time | 6 hours
  The procedure time is from skin cut to skin suture

CONTACTS AND LOCATIONS:
Overall Officials: Bentong Yu, MD, Study Director — 1st Affiliaed Hospital of Nanchang University
Locations (1):
- Surgery Building of 1st Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China